CLINICAL TRIAL: NCT04977843
Title: Effect of Early Bronchoalveolar Lavage on Severity of Ventilator Associated Pneumonia Assessed Through Clinical Pulmonary Infection Score on the Patients of Traumatic Brain Injury in Neurocritical Care.
Brief Title: Effect of E-BAL on Severity of VAP Assessed Through CPIS on the Patients of Traumatic Brain Injury in Neurocritical Care, Also Effect on Days of Ventilation and ICU Stay.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinnah Hospital (Other)
Responsible Party: Principal Investigator, Nazir Ahmed, medical officer trainee, Jinnah Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 62/erb
Record Dates: First submitted 2021-06-09; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Traumatic Brain Injury; Ventilator Associated Pneumonia
Keywords: Early Bronchoalveolar Lavage; CPIS
MeSH Terms: conditions — Brain Injuries, Traumatic; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- E-BAL (Experimental): E-BAL carried out within 48 hours
  Interventions: Procedure: EARLY BRONCHOALVEOLAR LAVAGE
- Conservative/Control (No Intervention): Standard of care management

INTERVENTIONS:
Procedure: EARLY BRONCHOALVEOLAR LAVAGE — E-BAL done with instillation of 100cc normal saline and sucked out
  Arms: E-BAL

SUMMARY:
Severe traumatic brain injury (STBI) is a leading cause of disability, mortality, and economic burden worldwide. The impact of severe traumatic brain injury (STBI) on the economy of developing countries like Pakistan is distressing. Pakistan has a large proportion of the young adult population in the World. Motorbike is the most common locomotive vehicle. These young ones are in the economically productive part of their lives. Their loss is an economical set back not only for their families but also for the Nation. Patients with STBI need standardized management in Neuro-critical care unit (NCCU). Although the setup and maintenance cost of an effective NCCU is one of the major burden on the budget of any public sector hospital, but the young survivor in turn can be productive for the Nation.

During mechanical ventilation, severe traumatic brain injury patients frequently develop ventilator-associated pneumonia (VAP). Ventilator-associated pneumonia can be evaluated using Clinical pulmonary infection score (CPIS). CPIS is considered as an important clinical indicator of pneumonia in NCCU.

Bronchoalveolar Lavage (BAL) is a minimally invasive procedure done with instillation of normal saline into subsegments of the lung followed by suction and collection of the instilled fluid for analysis with flexible bronchoscope. Patients with moderate and severe traumatic brain injury usually present with altered conscious level, and most of them already have aspiration of vomitus, debris and secretions which increase the risk of VAP in them. Bronchoalveolar lavage can be helpful in preventing this dreadful VAP by clearing the airways.

The aim of this study is to find out the effect of early Bronchoalveolar Lavage on severity of development of VAP assessed through clinical pulmonary infection score (CPIS) in TBI patients.

DETAILED DESCRIPTION:
Severe traumatic brain injury is a serious and ever growing issue of public health and the social economy of the World. It comprises 10% of all brain injuries and contributes to the high proportion of disabilities and deaths (McGarry et al., 2002; Mosenthal et al., 2002). STBI has a high mortality rate with prolonged hospital stay on average 17.5 days (Tagliaferri et al., 2006). The 14-day mortality on average remained 30.2%and most patients died in 48 hours (Braun CT, 2015). In the United States, approximately 235,000 patients were treated in the hospital per year due to traumatic brain injury (TBI). The estimated annual death rate in the US is about 50,000 cases per annum, with 21 to 400 billion US dollar annual costs due to TBI(Corrigan, Selassie and Orman, 2010; Marin, Weaver and Mannix, 2017). The annual cost of hospitalization due to traumatic brain injury (TBI) in China was 800 billion US dollars, with a mortality rate 9.8% (Liet al., 2015).

The complete recovery of a patient of STBI to pre-injury level is uncommon. Approximately 60% of the patient has ongoing impairment in the area of cognitive competency, gross motor activity, and recreational activity (Dikmen et al., 2003). Patients with STBI can have airway obstruction, aspiration, and hypoxia (Jovanovic et al., 2015). Mechanical ventilation is indicated in many patients with severe TBI(Jovanovic et al., 2015; Li et al., 2015). It maintains the oxygenation, protects airways, and maintains respiration. Most of the patients about 80% wean of early within 7 days from the mechanical ventilation without a respiratory problem, once the acute physiological disorder is corrected. However, 20% of patients still require prolonged mechanical ventilation after 7 days (Hess and MacIntyre, 2011). During the first four days, ventilator-associated pneumonia occurs in about 60% of the patients with severe traumatic brain injury (Ensault et al., 2017). The early systemic inflammatory response to head trauma patients predispose to early-onset VAP (Hedrick TL et al., 2008), while late-onset VAP that occurs after five days of mechanical ventilation (MV) is caused mainly by drug-resistant bacteria (Garnacho-Montero et al., 2014). Patients on mechanical ventilation have high morbidity, mortality, and infection rate due to acute respiratory distress syndrome and pulmonary embolism from venous thromboembolism (Nair and Niederman, 2015).

They also have decreased consciousness levels, disrupted natural defense barriers, decreased mobility, and lack of ability to protect the airways which can lead to pulmonary complications. Data is limited about effect of VAP in patients with STBI outcome. However multi organ failure has been identified as an independent contributor of poor outcomes in patients with severe TBI(Zygun et al., 2005).

A simple tool for the diagnosis of VAP was needed, thus a scoring system was developed in 1991, which included 7 clinical parameters for VAP diagnosis and it was named as Clinical Pulmonary Infection Score (CPIS) (Pugin J. Et al 1991) . The diagnosis of VAP was made using body temperature, leukocyte count and morphology, the character of tracheal secretion, PaO2 / FiO2 ratio, presence of pulmonary infiltration and its progression and microbiological culture results. A score of 6 or more suggests VAP (Basyigit. 2017).

Bronchoalveolar Lavage (BAL) is a minimally invasive procedure done with instillation of normal saline into subsegments of the lung followed by suction and collection of the instilled fluid for analysis. Loftus et al concluded in their study in 2017 that over half of all intubated patients with head or chest injury had evidence of pneumonia on Early Bronchoalveolar Lavage (E-BAL) performed within 48 hours of admission. E-BAL was associated with early discontinuation of antibiotics (7.3 vs 9.2 days), fewer days on mechanical ventilation (10.5 vs 16), fewer tracheostomies (49% vs 75%) and shorter ICU length of stay compared to L-BAL triggered by clinical suspicion of pneumonia (12 vs 17days). So, they found E-BAL useful for intubated patients with TBI or chest trauma. But the effect of this early lavage on severity of VAP assessed on CPIS is lacking. This study will help in determining the effect of early bronchoalveolar lavage on VAP in ventilated moderate and severe traumatic brain injury patients and will reflect the effect of early bronchoalveolar lavage on VAP through CPIS which can serve as prognostic indicator.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the age of 15-60 years with traumatic brain injury,
2. Presenting GCS between 5 to 10,
3. On mechanical ventilation,
4. Either gender.

Exclusion Criteria:

1. Patient undergoing neurosurgical procedure.
2. Poly trauma.
3. An underlying malignancy.
4. Patients admitted with any medical comorbidity including known case of restrictive or infiltrative lung disease, chronic liver disease, and chronic kidney failure.
5. Patients who expired within 10 days of admission.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
VAP severity | 10 days
  The study will help to figure out the effect of early bronchoalveolar lavage on decreasing the severity of VAP which will be assessed through CPIS
Ventilation Days | up to three weeks
  Number of days patient remains on ventilator
ICU stay Total | up to four weeks
  Number of days patient remains in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Syed S Hussain, MBBS, FCPS, Study Chair — Jinnah Hospital Lahore
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided